CLINICAL TRIAL: NCT00258128
Title: Effect of Salicylate on Glucose Metabolism in Insulin Resistance States
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CHS 00-01; R37DK051729 (NIH); R01DK051729 (NIH)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): This third small study has a randomized, masked, placebo controlled parallel design to compare salsalate 4.0 g/d to placebo. This is the salsalate 4.0 g/d arm.
  Interventions: Drug: Salsalate
- Placebo (Placebo Comparator): This third small study has a randomized, masked, placebo controlled parallel design to compare salsalate 4.0 g/d to placebo. This is the placebo arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salsalate — Active
  Other Names: Disalcid
  Arms: Treatment
Drug: Placebo — Placebo for salslate, used only in the third trial
  Arms: Placebo

SUMMARY:
Data supports diet induced obesity leads to activation of the IKK/NF-kB inflamatory pathway and that chronic inflammation leads to insulin resistance and diabetes. In rodents, salicylates inhibit IKK/NF-kB and may improve insulin sensitivity. We will study if this is true in people.

DETAILED DESCRIPTION:
Please see the following review articles on this topic:

Shoelson SE, Lee J, Goldfine AB. (2006) Inflammation in insulin resistance. J. Clin. Invest. 116, 1793-1801.

Goldfine AB, Fonseca V and Shoelson SE (2010) Therapeutic approaches to target inflammation in type 2 diabetes. Clin Chem. 57, 162-167.

Donath MY and Shoelson SE (2011) Type 2 diabetes as an inflammatory disease. Nat Rev Immunol. 11, 98-107.

Goldfine AB and Shoelson SE (2017) Therapeutic approaches targeting inflammation for diabetes and associated cardiovascular risk. J Clin Invest. 127, 83-93.

ELIGIBILITY:
Inclusion Criteria:

age 18 to 65 years, inclusive; HbA1c >6.0% (off medication-diabetic) normal hemoglobin and hematocrit, without donation of blood in the previous 2 months; without involvement in any study evaluating an investigational drug or device for the previous 2 months; normal clotting studies; female postmenopausal or surgically sterile, or using barrier or oral contraception and with a negative pregnancy test.

Exclusion Criteria:

pregnant or lactating women; patients with persistent ketonuria or a history of ketoacidosis (suggesting the need for insulin therapy); current of previous use of insulin for glucose control; patients with abnormal liver function defined as elevation of bilirubin, alkaline phosphatase, ALT, AST, or GGTP more than 1.5 times the upper limit of normal; patients with kidney disease (serum creatinine > 1.5 mg/dL) macroalbuminuria (1+ protein on a standard urine dip-stick, or > 300 mg urinary albumin/day)- (patients with microalbuminuria will be enrolled); patients with any significant diseases or conditions, including emotional or psychiatric disorders and substance abuse, including history of binge drinking, that, in the opinion of the investigator, are likely to alter the patient's ability to complete the study; patients with metabolic acidosis (abnormal anion gap); history of gastric ulcer, dyspepsia, or upper or lower GI bleed; history of allergy to aspirin, or bleeding diathesis or currently on oral anticoagulants including warfarin, heparin, aspirin or other NSAIDs; patients with major vascular event within 6 months of screening for the study (e.g., myocardial infarction stroke, coronary artery bypass graft (CABG) surgery, angioplasty, peripheral vascular surgery); patients with chronic heart disease, or a history of myocardial infarction or stroke. Symptomatic angina pectoris or cardiac insufficiency as defined by the NYHA; classification as Functional Class III or IV; patients with HbA1C > 13% (normal range 4-6%); patients who smoke more than one pack of cigarettes daily; patients taking treatment medications known to affect insulin sensitivity (e.g. diuretics, beta-blockers); patients taking warfarin, heparin or NSAID on a chronic basis; patients with inadequately controlled serum lipid levels (total cholesterol ≥ 275 mg/dL and fasting triglycerides ≥ 450 mg/dL); patients with history of cancer within 5 years prior to screening for the study other than basal cell carcinoma; active alcohol or other substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2000-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shoelson, Principal Investigator — Joslin Diabetes Center

REFERENCES:
- [Background] Fleischman A, Shoelson SE, Bernier R, Goldfine AB. Salsalate improves glycemia and inflammatory parameters in obese young adults. Diabetes Care. 2008 Feb;31(2):289-94. doi: 10.2337/dc07-1338. Epub 2007 Oct 24. PMID 17959861
- [Background] Shoelson SE, Lee J, Goldfine AB. Inflammation and insulin resistance. J Clin Invest. 2006 Jul;116(7):1793-801. doi: 10.1172/JCI29069. PMID 16823477
- [Result] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was active between 2000-2008. The location was an accademic clinic setting in the USA.
Pre-assignment Details: Subjects were instructed to monitor fasting blood glucose levels and with symptoms of hyperglycemia or hypoglycemia, and to avoid changing dietary or exercise habits.
Period: Overall Study
Arm/Group | Salsalate 4.0 g/d | Placebo
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This trial planned 8-9 participants per arm.
Groups:
- Salsalate: Randomized cohorts - Active
- Placebo: Randomized cohorts - Placebo
- Total: Total of all reporting groups
Arm/Group | Salsalate | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12) | 54 (8) | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Glucose
Description: fasting glucose
Time Frame: 4 weeks
Population: Receiving one dose of study drug and with measured value
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Placebo; Salsalate: Fasting glucose
Arm/Group | Placebo | Salsalate
Number analyzed (Participants) | 9 | 8
mmol/L | 7.1 (0.3) | 6.4 (0.3)

2. Secondary Outcome: Adiponectin
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Salsalate | Placebo
Number analyzed (Participants) | 8 | 9
mg/ml | 22.7 (2.5) | 10.6 (2.0)

ADVERSE EVENTS:
Time Frame: one month
Groups:
- Salsalate: Active Drug
- Placebo: Placebo - for salsalate
Arm/Group | Salsalate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

LIMITATIONS AND CAVEATS:
Small study size, sort duration of treatment, multiple endpoints.

See manuscript:

Goldfine AB, et al. Clin Transl Sci. 2008 May;1(1):36-43.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes